CLINICAL TRIAL: NCT05814653
Title: Evaluating the Feasibility of a Primary Care-based Treatment for Restrictive Eating Disorders in Children and Adolescents in the Health System
Brief Title: A Study to Evaluate Primary Care Treatment for Adolescent Eating Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jocelyn R. Lebow, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-011880; 1R34MH128296-01A1 (NIH)
Record Dates: First submitted 2023-02-03; First posted 2023-04-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Eating Disorders
Keywords: Children and Adolescents
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT-PC delivered by a primary care provider (Experimental): Subjects will receive up to 18 sessions of FBT-PC, delivered by a primary care provider, at their primary care clinic over 6 months.
  Interventions: Behavioral: Family Based Treatment-Primary Care
- Standard FBT (Active Comparator): Subjects will receive up to 18 session of FBT, delivered by a specialist mental health provider at Mayo Clinic in Rochester, MN over 6 months.
  Interventions: Behavioral: Family-Based Treatment

INTERVENTIONS:
Behavioral: Family Based Treatment-Primary Care — Novel treatment that borrows key intervention strategies from standard family-based treatment. It uses trained primary care providers (PCPs), in consultation with a mental health provider, to deliver family-based treatment strategies in community-based clinics to increase caregiver self-efficacy to reverse their child's dietary restriction and weight loss.
  Other Names: FBT-PC
  Arms: FBT-PC delivered by a primary care provider
Behavioral: Family-Based Treatment — Delivered by a mental health provider in a traditional mental health or eating disorder specialty setting. First-line evidence-based treatment for adolescent eating disorders that targets caregiver self-efficacy as a mechanism to facilitate weight restoration and ultimately symptom remission in adolescents.
  Other Names: FBT
  Arms: Standard FBT

SUMMARY:
The purpose of this study is to test the feasibility of a RCT of a new treatment for children and adolescents with eating disorders characterized by dietary restriction and/or weight loss or failure to gain expected weight. The treatment, which is called Family-Based Treatment for Primary Care (or FBT-PC for short), is based on Family-Based Treatment, the gold standard outpatient eating disorder treatment for children and adolescents.

DETAILED DESCRIPTION:
In the United States, half a million adolescents suffer from an eating disorder. With only 66 certified providers nationally, Family-Based Treatment (FBT), a first-line evidence-based treatment for adolescent eating disorders, is not readily available to most families. This provider shortage leaves most young patients without care and undoubtedly contributes to the chronicity and lethality of these conditions. Patients with eating disorders generally make their first contact with the healthcare system in primary care. As such, equipping primary care providers (PCPs) with effective means to treat these patients has potential to democratize care, improve rates of early intervention, and enhance patient outcomes. Family-Based Treatment for Primary Care (FBT-PC) is a novel intervention for delivery by a PCP in primary care that uses FBT strategies. Data support proof-of-concept for this adaptation. This study has several study aims. (1) Finalize the FB-PC intervention through an open case series. (2) Establish the feasibility and acceptability of FBT-PC for caregivers, patients, and PCPs in a pilot randomized controlled trial. Finally, (3) to test preliminary target engagement of FBT-PC and determine whether it is associated with improved caregiver self-efficacy and, through this mechanism, symptom remission. Remission will be defined as weight restoration to 95% of expected body weight and a score within 1 SD of community norms on the Eating Disorder Examination-Questionnaire. In addition, as (4) an exploratory aim analyses will be conducted to evaluate baseline characteristics of the sample to determine for whom the FBT-PC intervention is most beneficial. To accomplish all aims an open case series (n = 6) will be conducted, followed by a pilot trial in which 40 patients (ages 7-18 years) with restrictive eating disorders and their caregiver(s) will be randomly assigned to FBT-PC or a control condition of standard FBT. Families will attend up to 18 sessions over 6 months. Goals from the open case series (Aim 1) will include the development of tools for FBT-PC training and implementation, including treatment and training protocols and fidelity measures. Feasibility (Aim 2) will be assessed through an evaluation of recruitment and retention. Acceptability (Aim 2) will be evaluated using mixed methods surveys and interviews of caregivers, patients and PCPs on the topics of tolerability, fit, and burden. The degree to which FBT-PC engages the proposed mechanism of change, caregiver self-efficacy, to facilitate symptom remission will also be assessed (Aim 3). Effect sizes will be calculated for FBT-PC with a goal of ≥ 0.5, comparable with those found in FBT trials. Finally, baseline sample characteristics (Exploratory Aim) will be assessed including caregiver perceptions about their child's illness, referral method, length of illness, and symptom severity. Once feasibility, acceptability, and target engagement of the FBT-PC intervention have been established, these findings will be used in support of a large pragmatic clinical trial to evaluate the noninferiority of effectiveness of FBT-PC versus standard FBT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a DSM-5 restrictive eating disorder (anorexia nervosa or other specified feeding or eating disorder characterized by dietary restriction and/or weight loss or failure to make expected weight gains).
* Eligible patients will have at least one caregiver who is also willing to participate in the study.
* Eligible patients must receive primary care through the MCHS

Exclusion Criteria:

* Patients will be excluded who have received FBT in the past, and/or who report active suicidality.
* Patients who become physically or psychiatrically unstable during the study will be re-evaluated and referred for appropriate treatment.
* Patients will be excluded if their enrolled caregiver has active substance dependence, mental health concerns that make it difficult to engage in treatment, or are perpetrators of abuse.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment across 3 years | Rate of recruitment at end of study (3 years)
  Recruitment rate will be tracked, with a goal of enrollment of 75% of eligible participants.
Rate of retention across 3 years | Rate of retention at end of study (3 years)
  Retention rate will be tracked, with a target retention rate (attendance at >80% of sessions) of 70%.
Mixed methods feedback survey at end of treatment (caregiver/patient) | Assessed after the final session (within 6 months)
  This is a unique survey with quantitative (Likert scale rating/ yes/no questions) and qualitative (short answer) questions that assesses treatment satisfaction, acceptability of session frequency, length, and therapeutic alliance, as well as comfort and familiarity with treatment intervention components. Higher scores on Likert scales indicate greater satisfaction/acceptability.
Rate of retention across 3 years | Rate of retention at end of study (3 years)
  Rate of retention (defined as attendance at > 80% of sessions) will be tracked, with a target of <30% attrition.

SECONDARY OUTCOMES:
Parents versus Anorexia Scale (caregiver) | Monthly across the intervention (up to 6 months)
  The degree to which FBT-PC engages the proposed mechanism of change, caregiver self-efficacy, will be assessed through this well-validated caregiver-report measure. This is a 7-item of caregiver self-efficacy that has been widely used in the eating disorder treatment literature. Items assess parental efficacy in the Maudsley model of family-based treatment for anorexia nervosa. Scores range from 5-35, with higher scores indicated higher self efficacy
Parent Sense of Competency Scale (caregiver) | Monthly across the intervention (up to 6 months)
  The degree to which FBT-PC engages the proposed mechanism of change, caregiver self-efficacy, will be assessed through this well-validated caregiver-report measure, a 17-item measure of general parenting competency beliefs. Items are rated on a 1-6 Likert scale, with scores ranging from 17-102, with higher scores indicating higher parenting competency beliefs.
Eating Disorder Symptom Reduction (patient) | Pre/post intervention (up to 6 months)
  Patient weight restoration and reduction in behavioral/cognitive eating disorder symptoms as measured by the Eating Disorder Examination-Questionnaire or child Eating Disorder Examination-Questionnaire for patients ages 7-12. Higher scores on the 4 subscales and Global scale of these measures range from 0-6, with higher scores indicating more severe eating disorder symptomology.
Internalized Stigma of Mental Illness Scale (caregiver/patient) | Pre/post intervention (up to 6 months)
  The internalized stigma of having an eating disorder will be measured by the Internalized Stigma of Mental Illness Scale, a 20-item measure. This measure has been validated in populations of patients with eating disorders and will be modified to also be relevant for caregivers. Items are rated 1-4, with possible scores ranging from 29-116. Higher scores indicate higher internalized stigma.
Treatment experience feedback survey- Year 1 (provider) | End of Year 1 of the study
  Mixed methods surveys will be collected from primary care providers providing FBT-PC and within the participating practices, to assess their perceptions of their experience providing and referring to the intervention. HIgher scores on quantitative items (Likert scales rated 1-5) will indicated greater satisfaction.
Treatment experience feedback survey- Year 2 (provider) | End of Year 2 of the study
  Mixed methods surveys will be collected from primary care providers providing FBT-PC and within the participating practices, to assess their perceptions of their experience providing and referring to the intervention. HIgher scores on quantitative items (Likert scales rated 1-5) will indicated greater satisfaction.
Qualitative treatment experience feedback interview- Year 1 (provider) | End of Year 1 of the study
  30-60 minute semi-structured interviews will be conducted with primary care providers providing FBT-PC and within the participating practices, to assess their experience with the treatment (these will be open-ended qualitative questions)
Qualitative treatment experience feedback interview- Year 2 (provider) | End of Year 2 of the study
  30-60 minute semi-structured interviews will be conducted with primary care providers providing FBT-PC and within the participating practices, to assess their experience with the treatment (these will be open-ended qualitative questions)
Qualitative treatment experience feedback interview (caregiver) | At the end of their study participation (up to 6 months)
  Qualitative interviews will be conducted with a purposive combined sample of 10 caregivers from both arms, assessing their experience with both treatments and areas of ongoing need. These will be open-ended qualitative questions.
Qualitative treatment experience feedback interview (patient) | At the end of their study participation (up to 6 months)
  Qualitative interviews will be conducted with a purposive combined sample of 10 patients from both arms, assessing their experience with both treatments and areas of ongoing need. These will be open-ended qualitative questions.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Lebow, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials